CLINICAL TRIAL: NCT05174234
Title: Precariousness and Sexual Vulnerability During the Life Course and Migration of People From Haiti Living With or Without HIV in French Guiana (PARCOURS D'HAÏTI)
Brief Title: Precariousness and Sexual Vulnerability of People From Haiti Living With or Without HIV in French Guiana
Acronym: ParcoursHaiti
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: Parcours d'Haïti
Record Dates: First submitted 2021-10-25; First posted 2021-12-30 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: HIV Seropositivity
Keywords: hiv; haiti; french guiana; sexual health
MeSH Terms: conditions — HIV Seropositivity; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People living with HIV: a group of PLWHIV (n=400): women and men aged 18 to 60 years old from Haiti followed at the Cayenne Hospital, the Kourou Hospital or the West Guyanese Hospital (Saint Laurent du Maroni)
- People not living with HIV: a group of immigrants from Haiti not known to be infected with HIV (n=1600): women and men aged 18 to 60 years from Haiti
- People living with HBV: a group of PLWHBV (n=400): women and men aged 18 to 60 years old from Haiti followed at the Cayenne Hospital, the Kourou Hospital or the West Guyanese Hospital (Saint Laurent du Maroni)

SUMMARY:
French Guiana, a French territory located in South America, faces several social challenges including financial insecurity, unemployment and significant immigration. The degraded living conditions of migrants arriving in the territory are likely to put them in a situation of sexual vulnerability that could increase their risk of acquiring HIV (human immunodeficiency virus). This study proposes to conduct a survey of a group of people living with HIV in French Guiana who were born in Haiti and a group of Haitian people who are not HIV positive. With the help of interviewers who speak Haitian Creole, it will allow us to better understand the life paths of people from Haiti and their periods of vulnerability. Investigators will also focus on the use of testing and retention in care for those living with HIV. The results of this work will allow for the mobilization of resources and better adjustment of social support, prevention and care interventions implemented in French Guiana for migrant populations and/or those in precarious situations.

DETAILED DESCRIPTION:
French Guiana is a French overseas territory located in the Amazon basin of South America. It faces several challenges with dynamic demographics, poverty affecting nearly half of the population and significant immigration (more than a third of the Guianese population). People from Haiti represent 25% of foreigners living in French Guiana (census data, INSEE). This follows several waves of migration, including the major one dating from 2015. They are also over-represented among people living with HIV (PLWHIV). Work analyzing the slope of CD4 decrease and phylogeographic analyses suggests that a large proportion of HIV infections occur in French Guiana. The living conditions of Haitians after the arrival in French Guiana are often degraded, combining financial, administrative and housing precariousness. These conditions could increase the risk of having sex at risk of acquiring HIV and sexually transmitted infections when they occur in a context of social or sexual vulnerability or of priced intercourse in a context of survival. The 2013 ANRS-Parcours survey highlighted this sexual vulnerability among immigrants from sub-Saharan Africa living in Ile-de-France, using a biographical methodology which allowed comparing living conditions with the sexuality of people.

The present project proposes to set up a cross-sectional epidemiological and biographical study among PLWHIV from Haiti and people born in Haiti who declare not to be infected by HIV. The aim of the study will be to assess the frequency of unsafe sex (including forced sex) after the arrival in French Guiana of people from Haiti and their association with living conditions and the acquisition of HIV infection, year by year. It looks for better understand the living conditions of Haitians people after their arrival in French Guiana, to shed light on the use of screening and the determinants of late diagnoses, the delay in entering care but also the retention in care after the diagnosis, especially during the particular period of the Covid 19 epidemic. PLWHIV will also be offered a phylogenetic study to better understand HIV transmission.

Recruitment will focus on a group of PLWHIV from Haiti followed at the Cayenne, Kourou or Saint-Laurent du Maroni hospital and a group of people born in Haiti uninfected followed by general medicine, the health center for the poor (Permanence d'Accès aux Soins de Santé) or by the Prevention Health Center of French Red Cross in the municipalities of Cayenne, Matoury, Macouria or Kourou. Social, demographic and administrative data relating to the migratory journey, sexuality, the use of screening, the tools of diversified prevention, entry and retention in care will be collected. Part of the information will be collected each year since arriving in France using a biographical grid.

The results of this study are likely to improve the understanding of the situations of sexual vulnerability of immigrants from Haiti with a view to setting up a course in sexual health integrating an offer of screening and medicalized prevention to reduce the risk of HIV infection, STIs (sexually transmitted infections), unwanted sexual intercourse and unwanted pregnancies. They will articulate with the work already underway to develop a prevention and care offer directly within the informal settlements where a population mainly from Haiti lives.

It will also help to better understand the journey of Haitian PLWHIV after their diagnosis and produce information useful for the implementation of actions likely to prevent patients from being lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

For the 3 groups, patient :

* Born in Haiti, regardless of current nationality and date of arrival in France
* Aged between 18 and 60 years' old
* Arrived in French Guiana for more than 3 months
* Not opposed to participating in the study

For the HIV group

* Living with HIV and diagnosed for more than 3 months, regardless of their status regarding hepatitis B and C
* Be followed by one of the study's partner physicians in the hospitals of Cayenne, Kourou or Saint Laurent du Maroni

For the HBV group

* Living with HBV and diagnosed for more than 3 months, regardless of their status regarding HIV and hepatitis C
* Be followed by one of the study's partner physicians in the hospitals of Cayenne, Kourou or Saint Laurent du Maroni

For the non-HIV group

* Declared not to be infected with HIV, regardless of their status with respect to hepatitis B and C
* Being followed by one of the study's partner physicians or being recruited in the public space of one of the cities targeted by the study (Cayenne, Matoury, Rémire-Montjoly, Macouria, Kourou, Montsinery-Tonnegrande, Saint-Laurent-du-Maroni or Mana)

Exclusion Criteria:

* Unable to answer the interviewer in French or Haitian Creole
* Persons under guardianship or trusteeship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A group of PLWHIV and a group of people from Haïti not living with HIV
Sampling Method: Non-Probability Sample
Enrollment: 2189 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Frequency of unsafe sex | at inclusion
  Frequency of unsafe sex (including forced and paid sex) after arrival in French Guiana of people from Haiti and its association with their living conditions and acquisition of HIV infection

SECONDARY OUTCOMES:
the number of countries of residence | at inclusion
  the number of countries of residence during the lifetime and the duration of residence in each country, as well as access to health coverage and first screening in years of increased migration from Haiti
level of precariousness | at inclusion
  type of housing
level of precariousness | at inclusion
  type of resources
level of precariousness - right to stay | at inclusion
  right to stay
level of precariousness - health coverage | at inclusion
  type of health coverage
level of precariousness - use of STI screening | at inclusion
  use of HIV and HBV screening year after year after arrival in French Guiana
delay between arrival in French Guiana and the first screening for sexually transmitted infections (STIs) and HIV diagnosis for positive persons | at inclusion
  Identification of factors associated with earlier screening among the social indicators mentioned above
Attendance at preventive medicine facilities | at inclusion
  Attendance at preventive medicine facilities
delay between diagnosis and entry into care. | at inclusion
  Description of prolonged disruptions in care. Associated factors.
number of partners | at inclusion
  number of partners in the course of a lifetime and in the last twelve months, long relationships, occasional relationships, economic-sexual exchanges, forced relationships, recourse to paid sex year after year.
description of clades of the Pol gene of the HIV genotyping sequence | at inclusion
  list of clades of the Pol gene of the HIV genotyping sequence (Pol gene sequence) performed at the beginning of the care of participants living with HIV (phylogenetic analysis).
birth control methods used | at inclusion
  birth control methods used
number of desired and unwanted pregnancies | at inclusion
  number of desired and unwanted pregnancies
number of voluntary termination of pregnancy | at inclusion
  number of voluntary termination of pregnancy
number of abandonment of care during the Covid-19 epidemic | at inclusion
  number of abandonment of care during the Covid-19 epidemic
number in break in follow-up and treatment during the Covid-19 epidemic | at inclusion
  number in break in follow-up and treatment during the Covid-19 epidemic
delay in care during the Covid-19 epidemic | at inclusion
  delay in care during the Covid-19 epidemic

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MD Vignier, PhD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, France, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alcouffe L, Tareau MA, Brun Rambaud G, Lucarelli A, Boutrou M, Thorey C, Cantalupi G, Kpossou K, Huber F, Rabier S, Rochemont DR, Blaise T, Thomas E, Jean G, Pierre Louis R, Zephirin A, Basurko C, Djossou F, Cisse H, Faurous W, Drouaud Q, Mergeay-Fabre M, Adenis A, Nacher M, Vignier N. Sexual Health Determinants During the Life Course and Migration of Haitian-Origin People in French Guiana: Protocol for the Parcours d'Haiti Biographical and Transdisciplinary Study. JMIR Res Protoc. 2025 Jun 12;14:e63586. doi: 10.2196/63586. PMID 40505127